CLINICAL TRIAL: NCT06043934
Title: Effects of Neural Mobilization With and Without Intermittent Cervical Traction on Grip Strength, Sleep Quality, and Quality of Life in Cervical Radiculopathy
Brief Title: Neural Mobilization With Intermittent Cervical Traction on Grip Strength, Sleep Quality, and Quality of Life in Cervical Radiculopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Lahore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-UOL-507-08-2023
Record Dates: First submitted 2023-09-12; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Cervical Radiculopathy
Keywords: Cervical Radiculopathy; Pain; Sleep Quality; Quality of Life; Grip Strength; Intermittent Cervical Traction; Neural Mobilization
MeSH Terms: conditions — Radiculopathy; Pain; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neural Mobilization with Intermittent Cervical Traction (Experimental): Patients in this experimental group will receive neural mobilization with intermittent cervical traction and routine physical therapy.
  Interventions: Other: Neural Mobilization with Intermittent Cervical Traction
- Neural Mobilization (Active Comparator): Patients in this control group will receive neural mobilization and routine physical therapy.
  Interventions: Other: Neural Mobilization

INTERVENTIONS:
Other: Neural Mobilization with Intermittent Cervical Traction — This group will receive Neural Mobilization with Intermittent Cervical Traction along with routine physical therapy. The patient will be positioned in a supine position with 10 to 15 degrees of flexion on a comfortable treatment table. A suitable pillow will be arranged to support their head. The cervical traction device's integrity and readiness will be confirmed by the therapist. The starting weight will be about 10% of the patient's body weight, and this will slowly increase up to an appropriate level. The on-and-off times will be decided based on the patient's comfort and specific condition. Generally, a ratio of 3:1 or 4:1 (hold: rest) is used. For instance, 60 seconds of traction followed by 20 seconds of rest. The total treatment time will generally range between 15-20 minutes for 3 to 4 times per week. Participants will be scheduled to attend 12 treatment sessions ( 3-4 sessions every week for 4 weeks; 45 min each session).
  Arms: Neural Mobilization with Intermittent Cervical Traction
Other: Neural Mobilization — This Group will receive Neural Mobilization with routine physical therapy. Each nerve glide exercise will be performed ideally around 2-3 times, depending on the patient's comfort and tolerance levels. The intensity of the exercise is governed by the degree of stretch applied to the nerve. This should be within the patient's comfort level, causing a mild stretching sensation rather than pain. Each nerve glide will be performed in a set of 10-15 repetitions. Rest periods should be provided between each repetition and set, ensuring the patient's comfort.
  In median nerve glide the patient will be seated comfortably. Their arm will be guided into shoulder depression, elbow extension, forearm supination, and wrist and finger extension. The patient will then be instructed to slowly flex and extend their wrist while maintaining the other positions. Participants will be scheduled to attend 12 treatment sessions ( 3-4 sessions every week for 4 weeks; 45 min each session).
  Arms: Neural Mobilization

SUMMARY:
Cervical radiculopathy commonly called "pinched nerve," occurs when a nerve in the neck is compressed or irritated where it branches away from the spinal cord. This may cause pain that radiates into the shoulder and/or arm, as well as muscle weakness and numbness.

DETAILED DESCRIPTION:
Cervical radiculopathy (CR) is a disorder of the peripheral nervous system that affects the normal function of the cervical nerve roots (CNRs). It is frequently linked to chronic pain and daily functional limitations. The goal of the neural tissue mobilization technique is to restore the nervous system's capacity to tolerate the normal compressive, tensile, and frictional forces that are associated with day-to-day activities and to examine the neural tension in nerves and mobilize the nerves that exhibit neural tension through passive and active movements using tensioning and gliding. Cervical traction reduces pressure within the vertebral disks and unloads the structures of the spine by stretching muscles and ligaments. They are clinically important techniques that are easily understood by patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of any gender
2. Age between 35 and 55 years
3. Experience of unilateral upper-extremity pain, numbness, or paranesthesia. This must include a history of neck pain associated with radicular pain below the occiput and on one side of the neck, along with a tingling sensation on the lateral aspect of the elbow joint.
4. Positive results in at least three out of four tests Spurling's test, Distraction test, Upper Limb Neurodynamic Test 1, and ipsilateral cervical rotation of less than 60°, according to a clinical prediction rule.

Exclusion Criteria:

1. History of previous cervical or thoracic spine surgery
2. Bilateral upper-extremity symptoms
3. Signs or symptoms of upper motor neuron disease
4. Medical "red flags" (e.g. tumor, fracture, rheumatoid arthritis, osteoporosis, prolonged steroid use)

4. Injections in cervical spine in the past 2 weeks

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 85 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | Pain intensity will be measured at baseline, and change in pain intensity will be measured at 2nd week and 4th week of treatment session.
  Pain intensity is assessed using the Visual Analogue Scale (VAS), a unidimensional measure of pain intensity. The scale ranges from 0 (no pain) to 10 (worst possible pain), with the patient asked to rate their current level of pain.
Status of Sleep Quality | Sleep quality will be measured at baseline, and change in sleep quality status will be measured at 2nd week and 4th week of treatment session.
  Sleep quality is evaluated using the Chronic Pain Sleep Inventory (CPSI), a self- administered, a multidimensional questionnaire that assesses sleep disturbances related to chronic pain. Patients report their sleep-related difficulties on a scale of 0 to 100, where 0 represents never having sleep disturbances and 100 represents always having sleep disturbances.
Change in Quality of Life | Quality of life will be measured at baseline, and change in quality of life will be measured at 2nd week and 4th week of treatment session.
  Quality of Life (QOL) is assessed using the SF-36 questionnaire, a standard, validated instrument for measuring health-related quality of life. The SF-36 covers eight health domains: physical function, role limitations due to physical health, bodily pain, general health, vitality, social functioning, role limitations due to emotional problems, and mental health. Its score ranges from 0 to 100 with 0 representing poor quality of life and 100 representing good quality of life.
Change in Grip Strength | Grip Strength will be measured at baseline, and change in grip strength will be measured at 2nd week and 4th week of treatment session.
  Grip strength is evaluated using an isometric dynamometer, a device designed to assess the maximum isometric strength of the hand and forearm muscles. Grip strength for males range from 40 to 64 kg and for females from 20 to 38 kg

CONTACTS AND LOCATIONS:
Overall Officials: Umair Ahmad, PhD, Study Director — University of Lahore
Locations (1):
- The University of Lahore, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: After publication of manuscript.